CLINICAL TRIAL: NCT05536869
Title: Prospective Multicenter Study Comparing a Cohort of Women Having a Classic Caesarean to a Cohort of Women Having a FAUCS Caesarean
Brief Title: Study Comparing a Cohort of Women Having a Classic Caesarean to a Cohort of Women Having a FAUCS Caesarean (FAUCS)
Acronym: FAUCS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ramsay Générale de Santé (Other)
Collaborators: European Clinical Trial Experts Network (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2019-A01220-57
Record Dates: First submitted 2022-09-08; First posted 2022-09-13 (Actual); Last update posted 2022-09-15 (Actual); Status verified 2022-09

CONDITIONS: Cesarean Section; Dehiscence; Extra Peritoneal Caesarean Section
MeSH Terms: interventions — Cesarean Section

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patient with intraperitoneal caesarean section (Active Comparator)
  Interventions: Procedure: Caesarean
- patient with extraperitoneal caesarean section (Experimental): Faucs technique
  Interventions: Procedure: Caesarean

INTERVENTIONS:
Procedure: Caesarean — Two different caesarean section techniques : intra or extraperitoneal

SUMMARY:
The main objective of this study is to compare the time taken to obtain "street fitness" status for women after extraperitoneal cesarean section compared to women after a classic cesarean section.

ELIGIBILITY:
Inclusion Criteria:

* Patient scheduled for a caesarean between 38 and 42 weeks pregnant
* Patient aged between 18 and 42 years old
* Singleton
* Caesarean section with a theoretical operating time < 1 hour (without major complications)
* Patient affiliated to a social security scheme
* Patient having signed the free and informed consent.

Exclusion Criteria:

* BMI > 40
* High blood pressure treated intravenously
* Pre-existing diabetes in pregnancy
* Allergy to analgesics
* Prenatal depression
* Pathological insertion of the placenta (placenta previa or accreta).
* History of major pelvic or abdominal surgery (myomectomy, peritonitis) other than caesarean section or minor surgery.
* Addiction (drugs)
* Pre-existing psychiatric pathology leading to a risk of impaired judgment or behavior.
* Patient participating in another clinical study with a drug or medical device
* Protected patient: Adult under guardianship, curatorship or other legal protection, deprived of liberty by judicial or administrative decision
* Patient hospitalized without consent.

Ages: 18 Years to 42 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 72 (Estimated)
Dates: Start 2021-12-27 (Actual); Primary Completion 2022-09-27 (Estimated); Study Completion 2023-07-27 (Estimated)

PRIMARY OUTCOMES:
The postoperative time in hours from which the patient stably fulfills the criteria for "street fitness". | 1 month
  These criteria are defined in the Chung score. This score is between 0 and 10 and evaluate the vital signs, wandering, nausea or vomits, pain and surgical bleeding.

CONTACTS AND LOCATIONS:
Locations (1):
- Les Franciscaines Clinic, Versailles, IDF, France